CLINICAL TRIAL: NCT01010087
Title: A Randomized, Double-Blinded Controlled Trial Comparing High vs Standard Dose Oseltamivir in Severe, Influenza Infection in ICU. "ROSII Study"
Brief Title: Trial Comparing High Versus Standard Dose Oseltamivir in Severe Influenza Infection in ICU
Acronym: ROSII
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Patient population no longer available.
Sponsor: University of Manitoba (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Anand Kumar MD, Winnipeg Regional Health Authority; Health Sciences Centre
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 133312
Record Dates: First submitted 2009-11-05; First posted 2009-11-09 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Influenza A Virus
Keywords: patients admitted to ICU
MeSH Terms: interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Oseltamivir dose 75 mg bid (Active Comparator): Standard dosing
  Interventions: Drug: Oseltamivir
- High Dose Oseltamivir arm 225mg bid (Experimental): High dose arm of the study
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Oseltamivir — standard (75 mg bid) or high-dose (225 mg bid) oseltamivir
  Other Names: Tamiflu

SUMMARY:
Primary Objectives:

The primary objective of the trial is to compare the antiviral efficacy of a 10 day course of standard (75 mg bid) and high-dose (225 mg bid) oseltamivir (or equivalent doses in mild-moderate renal failure) in the treatment of severe influenza infections.

The hypothesis is that high dose oseltamivir will increase the proportion of patients with negative reverse transcriptase (RT)-PCR detection of influenza viral RNA (and viral culture, at selected sites) at Day 5 post-treatment.

An important secondary objective of the trial, which reflects the main clinical objective, is to determine the difference in the numbers of ventilator days between the standard-dose and high-dose groups

DETAILED DESCRIPTION:
Primary Objectives:

The primary objective of the trial is to compare the antiviral efficacy of a 10 day course of standard (75 mg bid) and high-dose (225 mg bid) oseltamivir (or equivalent doses in mild-moderate renal failure) in the treatment of severe influenza infections.

The hypothesis is that high dose oseltamivir will increase the proportion of patients with negative reverse transcriptase (RT)-PCR detection of influenza viral RNA (and viral culture, at selected sites) at Day 5 post-treatment.

An important secondary objective of the trial, which reflects the main clinical objective, is to determine the difference in the numbers of ventilator days between the standard-dose and high-dose groups.

Secondary Objectives:

* Laboratory objectives:

  1. Assess viral RNA load and clearance from nasopharyngeal and tracheal aspirate (intubated) or oropharyngeal (non-intubated) samples by RT-PCR on days 1, 3, 5, 7, 10, 14 and 28 days
  2. Determine viral clearance by culture from nasopharyngeal and tracheal aspirate (intubated) or oropharyngeal (non-intubated) samples on days 1, 3, 5, 7, 10, 14 and 28 days at select hospital sites with culture capability
  3. Assess the pharmacokinetics of oseltamivir carboxylate and phosphate on Day 3 in suspected H1N1 patients with respiratory distress and/or critical illness requiring ICU care
  4. Characterize the inflammatory cytokine response on Day 1-3, 5, 7, 10, 14, 21 and 28 days to severe influenza stratified by standard-dose versus high-dose oseltamivir therapy.
  5. Assess leukocyte gene expression at day 1, 3, 5, 10 and 21 days using high throughput RNA assessment techniques
  6. Examine urine for biomarkers of disease and severe disease
* Clinical and Safety Objectives:

  1. Determine the difference in the number of ventilator days in the standard-dose and high-dose groups
  2. Determine tolerability of high-dose versus standard-dose oseltamivir as assessed by the number of serious, atypical and drug-related adverse events that are possibly or probably related to oseltamivir
  3. Assess other secondary efficacy variables including survival duration, hospital free days to day 60, ICU free days to day 60, and shock (ie vasopressor) and renal failure free (ie not requiring hemodialysis; ultrafiltration acceptable) days to day 28 in relation to high vs standard dose oseltamivir therapy
  4. Assess 60 day mechanical ventilation and ICU-free days stay in relation to high vs standard dose oseltamivir therapy
  5. Determine clinical criteria used by clinicians when electing to continue or re-initiate oseltamivir therapy beyond 10 study day treatment course

Tertiary Objectives: Exploratory Analyses

* Laboratory Objectives:

  1. Assess the relationship between pharmacokinetic variables on day 3 and measures of viral clearance
  2. Assess the frequency and genetic basis of antiviral resistance to oseltamivir during and after therapy
  3. Determine possible host genetic factors including HLA type that predispose to severe influenza
* Clinical and Safety Objectives:

  1. Determine differences in development and persistence of adverse clinical signs (fever, heart rate, hypotension), requirement for and duration of organ support (supplemental oxygen, vasopressor/inotropes, continuous renal replacement therapy) and occurrence and resolution of organ failure by Sequential Organ Failure Assessment (SOFA) score at days 7, 10, 14 and 28 as a consequence of high-dose versus standard-dose oseltamivir
  2. Determine impact of oseltamivir dosing on frequency of progression to mechanical ventilation among non-ventilated patients

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 12 and older and 45 kg or more
2. Suspected or confirmed influenza (Appendix A)
3. Requirement for ICU admission due to respiratory distress or critical illness defined as one of:

   1. Inspired oxygen need of >50% for at least 4 hours (For FiO2 for non-intubated patients see Appendix B)
   2. mechanical ventilation
   3. Patient is receiving inotrope or vasopressor
4. Negative b-HCG test or negative bedside urine test pending a confirmatory b-HCG test for pregnancy in women of childbearing age (12-60 years of age) will allow study entry

Exclusion Criteria:

1. Inability to obtain consent
2. Patients receiving more than two doses of 150 mg or higher oseltamivir in 36 hours before study entry
3. Patients having received more than 3 doses of 75 mg oseltamivir immediately in 36 hours before study entry
4. Age less than 12 years, or age <16 and weight less than 45 kg
5. Unlikely to absorb enteral study drug (e.g. patients with partial or complete mechanical bowel obstruction, intestinal ischemia, infarction, and short bowel syndrome)
6. Known allergy or hypersensitivity to oseltamivir
7. Pregnancy or breast feeding
8. Previous enrollment in current study
9. Concurrent involvement in an RCT examining an antiviral agent including other neuraminidase inhibitors, interferon-a and/or ribavirin
10. Chronic renal failure requiring chronic hemodialysis
11. Severe chronic liver disease (Child-Pugh Score 11-15)
12. Anticipated death within 24 hours as judged by attending physician or local PI
13. Patient carrying "do not intubate" order (a "no CPR" or "no defibrillate" or "no chest compressions" order alone is allowed)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Negative reverse transcriptase (RT)-PCR detection of viral RNA in nasopharyngeal and tracheal aspirate (intubated) or oropharyngeal (non-intubated) samples at Day 5 among patients who require ICU admission due to respiratory distress. | Day 5 on study

SECONDARY OUTCOMES:
Ventilator days up to 60 d (main clinical endpoint), | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Anand Kumar, MD, Principal Investigator — University of Manitoba
Locations (1):
- Winnipeg Regional Health Authority; Health Sciences Centre, Winnipeg, Manitoba, Canada